CLINICAL TRIAL: NCT04123730
Title: Automated Oxygen Titration With O2matic During Walking in Patients With COPD
Brief Title: Automated Oxygen Titration During Walking in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Region Örebro County (Other); Aalborg University Hospital (Other); Danmarks Lungeforening (Other)
Responsible Party: Principal Investigator, Linette Marie Kofod, Physiotherapist, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-19044780
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Respiratory Failure
Keywords: Long Term Oxygen Treatment; Dyspnea; Physiotherapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency; Dyspnea

STUDY DESIGN:
Intervention Model Description: randomised crossover trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient will be blinded for the oxygen supply. An independent person will prepare the oxygen setup with O2matic in manual mode for fixed dose oxygen and in automatic mode for automated oxygen titration. The assessor conducting the walking test is blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed dose oxygen (Active Comparator): O2Matic deliver the usual fixed-dose oxygen treatment during walking.
  Interventions: Other: Fixed-dose compared to variable oxygen flow supplementation during walking
- Automated oxygen titration (Experimental): O2Matic deliver a variable oxygen dosage set at an SpO2-target of 90 to 94 % and a O2-flow of 0 - 15 liters/min during walking.
  Interventions: Other: Fixed-dose compared to variable oxygen flow supplementation during walking

INTERVENTIONS:
Other: Fixed-dose compared to variable oxygen flow supplementation during walking — At day 1 the patients will perform Walk A and Walk B in a random order:
  Walk A: The patients will perform a Endurance Shuttle Walk Tests (ESWT) with the fixed-dose (FOT). O2matic will monitor pulse rate and saturation continuously during the test.
  Walk B: The patients will perform a Endurance Shuttle Walk Tests (ESWT) with a variable oxygen flow (AOT) depending on the saturation. O2matic will monitor pulse rate and saturation continuously during the test, and adjust oxygen flow depending on the saturation.
  At day 2 the patients will perform two 6 minutes walking (MWT) test in random order:
  Walk C: A 6 MWT with FOT Walk D; A 6 MWT with AOT

SUMMARY:
Purpose: to evaluate the immediate effect of automated oxygen titration compared to usual fixed-dose oxygen treatment during exercise in patients with COPD on long-term oxygen treatment.

Methods: The study will be conducted as a double blinded randomized crossover trial with two arms. 40 ambulatory patients with COPD and home oxygen treatment will be included from AHH Hospital's catchment area. The patients will conduct two Endurance Shuttle Walk Tests (ESWT) in a crossover design using an O2matic device to deliver a variable oxygen dosage set at an SpO2-target of 90-94% and an O2-flow of 0 - 15 liters/min and using the patients´ usual fixed-dose oxygen delivery, in a randomized order. In both arms O2matic will monitor pulse rate and SpO2 continuously during the test, but only in the automated oxygen titration arm will O2matic adjust oxygen flow. The patient and the physiotherapist supervising the tests will be blinded to the oxygen dose. Primary outcome is the changes in perceived dyspnea intensity using Borg CR10 scale between walking with automated titration compared to fixed-dose treatment. Secondary outcomes are differences in walking time, the average oxygen consumption between automated oxygen titration and fixed-dose treatment and difference in time spent within acceptable SpO2-interval.

DETAILED DESCRIPTION:
Long-term oxygen treatment (LTOT) at home is essential for patients with COPD and chronic hypoxemia. It is recommended that the given oxygen flow rate should be enough to keep the blood saturation (SpO2) between 90% and 94%. Although the oxygen need increases with activity, there is no consensus on oxygen dosage during activity (BTS-guideline).

The purpose of this study is to evaluate the immediate effect of automated oxygen titration (AOT) compared to usual fixed-dose oxygen treatment (FOT) during exercise in patients with COPD on long-term oxygen treatment.

Method The study will be performed on 40 patients with COPD and on LTOT. An incremental shuttle walk test (ISWT) will be performed to establish the walking speed corresponding to 75% of the estimated peak oxygen consumption. The patients will all use a rollator as walking aid and the oxygen equipment will be placed in the rollator. The patients will after inclusion conduct two Endurance Shuttle Walk Tests (ESWT) with FOT and AOT respectively in a randomized order. One ESWT will be performed using O2matic to deliver a variable oxygen dosage set at an SpO2-target of 90 to 94 % and a O2-flow of 0 - 15 liters/min (AOT). The other ESWT will be performed using the usual fixed-dose oxygen delivery (FOT).

The patients will also conduct two six minutes walking tests (6 MWT) with FOT and AOT in random order in the same way as mentioned above.

Assessments:

Demographic data, including body mass index, and smoking history, will be registered. Use of a rollator, and usual flow of oxygen supplementation will be registered. The score in the CAT- questionnaire (COPD Assessment Test, range of 0-40) will be registered along with the results of the MRC (Medical Research Council, range 1-5).

A lung function test will be performed using Medikro Pro Spirometer. Forced Expiratory Volume in the first second (FEV1) and Forced Vital Capacity (FVC) will be recorded. All lung function measures will be expressed in absolute values and in percent of predicted.

Dyspnea will be registered using Borg Dyspnea Scale CR10 (6). Before, and after completing the 6MWT the patients will be asked to rate their intensity of dyspnea. At the ESWT the patients will rate their intensity of dyspnea before and after completing the test and every minute during the test.

Hand grip strength will be measured using static hand squeeze around a dynamometer.

Walking tests:

Shuttle Walk Test will be performed using the Incremental Shuttle Walk Test (ISWT) followed by the Endurance Shuttle Walk Test (ESWT) on two different days. ISWT is initially conducted once for familiarization followed by a second test. The patients will be given a rest of 20 minutes between tests and the best result is recorded. The results of ISWT will be used to calculate the walking speed in the ESWT, which will be set at 75% of max and not 85% of max as the intension is to keep the patients walking for more than just 1-3 minutes. The patient is in both tests required to walk around two cones set 9 meters apart (so the final track is 10 meters). In the ESWT the patients are asked to walk as long as possible until they are unable to continue. The time walked in the ESWT will be registered.

The six-minute walking test (6 MWT), assesses the distance walked in metres over six minutes as a sub-maximal test of aerobic capacity/endurance. It requires the patient to walk between cones set 30 meters apart(8).

Walking limitation will be noted. The patients will be asked to report the primary limitation for not being able to walk longer: dyspnea, leg fatigue, pain, discomfort, anxiety or "other reasons".

Oxygen consumption and oxygen saturation (SpO2) will be registered using O2matic, a device which adjusts the oxygen flow to maintain the saturation within a target interval. O2matic is a device, which based on continuous, non-invasive measurement of SpO2 adjusts oxygen flow to the patient within a defined target interval. SpO2-target can be set individually, but in this study will be fixed at 90 to 94 %. If SpO2 falls below 90 % oxygen flow will increase, and if SpO2 increases above 94 % oxygen flow will decrease. The adjustments are done every second based on average SpO2 for the last 15 seconds. In case of low SpO2 (below target or below 85 %), low pulse rate (<45) or high pulse rate (user defined) an alarm will be visible and audible.

Statistical considerations and strength calculation:

The primary outcome is change in the BORG CR10 dyspnea scale. The minimal clinical important difference (MCID) is 1 unit (9) and standard deviation expected to be 2.0. Based on alfa of 0,05 and a power of 80 % a sample of 33 patients is needed to examine if AOT results in improvement in time walked during the ESWT. Due to possible dropout 40 patients will be included in the study. Categorical variables are compared using Chi-Square or Fisher's exact test, as appropriate. Continuous variables are examined for normality and analyzed with either unpaired t-test (in case of normality) or Wilcoxon-Mann-Whitney test (in case of non-normality). The Statistical Package SPSS ver. 22 will be used for all statistical analyses.

The study will take place at Hvidovre Hospital from October 2019 and until all 40 patients are included. Linette Marie Kofod is the principal investigator. The study will be conducted as an interdisciplinary collaboration between the Pulmonary Section and the Department of Physiotherapy, Amager and Hvidovre University Hospital, which have approved the study.

ELIGIBILITY:
Inclusion Criteria:

* Verified history of COPD with FEV1/FVC < 0,70
* Hypoxemic at rest (SpO2 ≤ 90 %) and fulfilment of criteria for LTOT
* Able to walk at least 70 meters
* Cognitively able to participate in the study and willing to give informed consent

Exclusion Criteria:

* Pulmonary or cardiac condition other than COPD limiting exercise performance
* Unstable heart condition or stenotic aortic valve disease
* A physical condition including paralysis, lower extremity pain, or back problem limiting exercise performance
* Exacerbation in COPD treated with either antibiotics or prednisolone within the last 3 weeks

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Perceived dyspnea intensity using Borg CR10 dyspnea scale | Twenty minutes
  Difference in Dyspnea Borg CR10 (from 0-10) scores in the ESWT at isotimes (every minute) in both tests walking with automated titration compared to fixed-dose treatment. The Borg scale starts at number 0 where your breathing is causing the patient no difficulty at all and progresses through to number 10 where the breathing difficulty is maximal

SECONDARY OUTCOMES:
Walking time | Twenty minutes
  Difference in walking time in minutes and seconds between groups in ESWT
Time with Hypoxemia | Twenty minutes
  Difference between groups in time spent within acceptable SpO2-interval (SpO2 90 - 94 %) and time spent with moderate hypoxemia (SpO2 < 88 %) and severe hypoxemia (SpO2 < 85 %).
Average numbers of liter oxygen per minutes | Twenty minutes
  Difference in average oxygen consumption between groups, measured with number of liter oxygen per minutes using O2Matic
Walking distance in meters | six minutes
  Difference in walking distance in meters between groups in 6 MWT

CONTACTS AND LOCATIONS:
Overall Officials: Linette Marie Kofod, PT, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Copenhagen University Hospital, Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. Data access in Denmark are under very strict juristic data protection law. Any possible access or sharing demands a part application to; (1) Danish Data Protection Agency, (2) Ethics Committee of the Capital Region, (3) National Health Data Authorities.
  Only if the applications are approved data will be considered available for sharing.
  The authors will not be able to support this process and a prolonged process must be expected
Supporting Information: Study Protocol, ICF
Time Frame: 01.01.2023
Access Criteria: Se Plan Description

REFERENCES:
- [Background] O'Driscoll BR, Howard LS, Earis J, Mak V; British Thoracic Society Emergency Oxygen Guideline Group; BTS Emergency Oxygen Guideline Development Group. BTS guideline for oxygen use in adults in healthcare and emergency settings. Thorax. 2017 Jun;72(Suppl 1):ii1-ii90. doi: 10.1136/thoraxjnl-2016-209729. No abstract available. PMID 28507176
- [Background] Hansen EF, Hove JD, Bech CS, Jensen JS, Kallemose T, Vestbo J. Automated oxygen control with O2matic(R) during admission with exacerbation of COPD. Int J Chron Obstruct Pulmon Dis. 2018 Dec 14;13:3997-4003. doi: 10.2147/COPD.S183762. eCollection 2018. PMID 30587955